CLINICAL TRIAL: NCT02145429
Title: Preventing Depression in Late Life: A Model for Low and Middle Income Countries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Goa Medical College (Other); Sangath (Other)
Responsible Party: Principal Investigator, Charles Reynolds, Professor in Geriatric Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R34MH096997-01A1 (NIH)
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Results first posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Depression; Anxiety Disorder
Keywords: Prevention of depression and anxiety disorder; Depression Prevention
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- problem solving therapy + Behavioral Treatment of Insomnia (Experimental): Problem Solving Therapy + Brief Behavioral Treatment of Insomnia as needed
  Interventions: Behavioral: Problem Solving therapy and Brief Behavioral Treatment of Insomnia
- Enhanced Usual Care (No Intervention): Care as usual with scheduled assessments of clinical status

INTERVENTIONS:
Behavioral: Problem Solving therapy and Brief Behavioral Treatment of Insomnia — Problem Solving therapy teaches problem solving skills that participants can use in their everyday life. A problem is identified, various solutions identified and explored with the underlying focus to learn behavioral and self management strategies.Social casework and management of chronic disease is also included as per the participant's need.
  Brief Behavioral Treatment of Insomnia focuses on improving sleep by promoting sleep hygiene such as time spent in bed and decreasing night time stimuli. The therapy has been suitably modified to suit the needs of the participants to be recruited in the Low and Middle income countries keeping in mind the low level of literacy and the local social and health care services.
  Arms: problem solving therapy + Behavioral Treatment of Insomnia

SUMMARY:
This study is being conducted in GOA India. The study addresses specific issues of depression prevention in older adults living in low- and middle income countries (LMICs), by developing risk-reduction strategies through the use of lay health counselors. We will be training Lay Health Counselors (LHC's) to deliver simple behaviorally oriented interventions, designed to enhance the ability to relax, to improve active coping via better problem solving, and to increase protective factors such as good quality sleep. Lay Health Counselors are inhabitants of Goa.

The aim of phase 1 is to create a depression and anxiety prevention intervention for use by lay health counselors. We will test the feasibility and acceptability of Problem Solving Therapy for Primary Care (PST-PC) and Brief Behavioral Treatment for Insomnia (BBTI). The products of phase 1 will be a prevention and counseling manual to standardize the implementation of the interventions for further testing in a randomized prevention trial (Specific Aim 2) and the adaptation of PST-PC and BBTI for the Indian population.

In Phase 2, we will: gather data on the feasibility of identifying, enrolling, randomizing and retaining participants; implement the experimental intervention and enhanced usual care; identify "real world", barriers and develop strategies for addressing them; and assess the fidelity of the interventions.

DETAILED DESCRIPTION:
Prevention of common mental disorders in older adults (major depression and anxiety disorders) in Low and Middle Income Countries (LMICs) is a major challenge in global mental health research. The public health imperative for devising strategies to prevent late life depression and anxiety in LMICs includes the rapid demographic transition and aging in countries like India, increased exposure of older adults to risk factors for depression (disability, depletion of economic and social resources, bereavement, care giving, and chronic insomnia), and workforce issues (such as a dearth of mental health specialists). The dearth of specialist resources, together with the limited ability of current depression treatments to avert years lived with disability, underscores the need for preventive interventions that can be delivered by lay health workers in non-health care or primary care settings. Such development could also benefit policy and practice in the US by clarifying appropriate roles for lay and non-specialist workers in depression and anxiety prevention for populations with few mental health resources. We propose to build upon the MANAS trial conducted in Goa, India. Given the shortage of mental health specialists in Low and Middle Income Countries (LMICs), MANAS (which means "project to promote mental health" in the Konkani language) employed the strategy of task-shifting, that is, the rational redistribution of tasks among health workforce teams to make more efficient use of lay human resources for health. MANAS demonstrated that the use of lay health counselors (LHCs), as part of a collaborative stepped care intervention, increases rates of recovery from common mental disorders (depression and anxiety) in public primary care facilities. In addition, preliminary evidence indicated that the MANAS model of using Lay Health Counselors in a stepped-care collaborative intervention may also reduce the incidence of common mental disorders in those who initially present with subthreshold (subsyndromal) depressive and anxiety symptoms. We propose to investigate translation of depression and anxiety prevention strategies to LMICs through non-specialist delivery systems. The goal of this study is to develop and pilot test in Goa, India a Lay Health Counselor-led depression and anxiety disorder prevention strategy, building upon the experience of the MANAS treatment trial called the DIL (Depression in Late Life) intervention.

Specific Aim (1) formative research (months 1 - 12): following Medical Research Council Guidelines for the development of complex interventions, we will create and standardize a MANAS-derived depression and anxiety prevention intervention (DIL Intervention) for use by lay health counselors (LHCs) in primary care clinics in Goa. We will develop an intervention manual based on the original MANAS trial and best practices for depression and anxiety prevention from the global literature. Via systematic study of an uncontrolled case series (enrolling 20 subjects), we will test the feasibility and acceptability of DIL Intervention. The DIL Intervention will comprise psychoeducational interventions delivered by Lay Health Counselors and previously shown to have prevention, such as Problem Solving Therapy for Primary Care (PST-PC) and Brief Behavioral Treatment for Insomnia (BBTI). The products of Specific Aim (1) will be a prevention manual to standardize the implementation of DIL Intervention for further testing in a pilot randomized prevention trial (Specific Aim 2), together with recruitment and assessment protocols and a randomization procedure.

Specific Aim (2) pilot randomized prevention trial (months 13 - 36): Via the use of a pilot randomized prevention trial (DIL Intervention) we will: gather data on the feasibility of identifying, enrolling, randomizing and retaining participants; implement the experimental intervention and enhanced usual care; identify "real world", barriers and develop strategies for addressing them; and assess the fidelity of the DIL implementation. As recommended in the R34 program announcement (PAR-09-173), we will collect measures of feasibility, acceptability, tolerability, and safety, rather than conducting formal tests of outcome or attempting to obtain an estimate of an effect size (because estimates are likely to be inflated and unstable.) These data will be critical to a subsequent confirmatory randomized depression prevention trial based in Goa and to our long-term goal of scalable depression prevention in Low and Middle Income Countries (LMICs).

ELIGIBILITY:
Inclusion Criteria:

* Patient at the participating primary care centers
* age 60 and older
* GHQ scores 4 or above
* Hindi MMSE scores 24 or higher
* no episodes of major depression or anxiety disorder within the past 12 months
* no current antidepressant pharmacotherapy

Exclusion Criteria:

* episode of major depression or anxiety disorder within the past 12 months
* current antidepressant pharmacotherapy
* younger than age 60
* Hindi MMSE scores less than 24
* GHQ scores less than 4

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles F Reynolds, MD, Principal Investigator — University of Pittsburgh; Amit Dias, MD, Principal Investigator — Sangath and Goa College of Medicine; Vikram Patel, MD, PHD, Principal Investigator — Sangath; Alex Cohen, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Goa Medical College, Bambolim, Goa, India

REFERENCES:
- [Derived] Dias A, Azariah F, Anderson SJ, Sequeira M, Cohen A, Morse JQ, Cuijpers P, Patel V, Reynolds CF 3rd. Effect of a Lay Counselor Intervention on Prevention of Major Depression in Older Adults Living in Low- and Middle-Income Countries: A Randomized Clinical Trial. JAMA Psychiatry. 2019 Jan 1;76(1):13-20. doi: 10.1001/jamapsychiatry.2018.3048. PMID 30422259

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Because enrollment exceeded expectations, we were able to increase sample size from the original n proposed (120) to 181, thereby allowing us to carry out a fully powered confirmatory RCT. We obtained NIMH permission to change from an intervention development study to an RCT
Groups:
- Problem Solving Therapy + Behavioral Treatment of Insomnia: Problem Solving Therapy + Brief Behavioral Treatment of Insomnia as needed
  Problem Solving therapy and Brief Behavioral Treatment of Insomnia: Problem Solving therapy teaches problem solving skills that participants can use in their everyday life. A problem is identified, various solutions identified and explored with the underlying focus to learn behavioral and self management strategies.Social casework and management of chronic disease is also included as per the participant's need.
  Brief Behavioral Treatment of Insomnia focuses on improving sleep by promoting sleep hygiene such as time spent in bed and decreasing night time stimuli. The therapy has been suitably modified to suit the needs of the participants to be recruited in the Low and Middle income countries keeping in mind the low level of literacy and the local social and health care services.
Period: Overall Study
Arm/Group | Problem Solving Therapy + Behavioral Treatment of Insomnia | Enhanced Usual Care
Started | 91 | 90
Completed | 75 | 79
Not Completed | 16 | 11
Not completed — Death | 4 | 5
Not completed — Lost to Follow-up | 4 | 3
Not completed — Withdrawal by Subject | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Problem Solving Therapy + Behavioral Treatment of Insomnia | Enhanced Usual Care | Total
Number analyzed (Participants) | 91 | 90 | 181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 91 | 90 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (7.1) | 69.7 (7.3) | 69.6 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 57 | 114
  Male | 34 | 33 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 91 | 90 | 181
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — All participants were recruited from Goa, India
  Participants
    India | 91 | 90 | 181

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Develop Major Depression and Anxiety Disorders
Description: Cumulative incidence of episodes of major depression and anxiety disorders over a 12-month period measured by MINI
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | Problem Solving Therapy + Behavioral Treatment of Insomnia | Enhanced Usual Care
Number analyzed (Participants) | 75 | 79
Participants | 4 | 13
Statistical Analysis 1: Comparison: Problem Solving Therapy + Behavioral Treatment of Insomnia vs Enhanced Usual Care; Test type: Other; p = 0.04, Log Rank; Hazard Ratio (HR) = 0.32, 95% CI 2-sided [0.10 to 0.98]

2. Primary Outcome: General Health Questionnaire (GHQ) Scores
Description: Levels of depressive and anxiety symptoms. Scores on the General Health Questionnaire (GHQ-12) range from 0 to 12; a higher score indicated greater symptoms for depression and anxiety
Time Frame: One year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Problem Solving Therapy + Behavioral Treatment of Insomnia | Enhanced Usual Care
Number analyzed (Participants) | 75 | 79
score on a scale | 3.67 (2.67) | 5.67 (3.19)
Statistical Analysis 1: Comparison: Problem Solving Therapy + Behavioral Treatment of Insomnia vs Enhanced Usual Care; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.18, 95% CI 2-sided [-2.03 to -0.31]

3. Secondary Outcome: World Health Organization Disability Assessment Schedule (WHODAS-II) Scores
Description: Assessment instrument for health and disability or functional status. Scores on the World Health Organization Disability Assessment Schedule (WHODAS 2.0) range from 12 to 60; a higher score indicated greater disability.
Time Frame: One year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Problem Solving Therapy + Behavioral Treatment of Insomnia | Enhanced Usual Care
Number analyzed (Participants) | 75 | 79
score on a scale | 16.72 (5.71) | 17.73 (6.27)
Statistical Analysis 1: Comparison: Problem Solving Therapy + Behavioral Treatment of Insomnia vs Enhanced Usual Care; Test type: Other; p = 0.26, Mixed Models Analysis; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-1.89 to 1.62]

ADVERSE EVENTS:
Time Frame: One Year
Arm/Group | Problem Solving Therapy + Behavioral Treatment of Insomnia | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 4/91 | 5/90
Serious Adverse Events (participants affected / at risk) | 19/91 | 5/90
Other Adverse Events (participants affected / at risk) | 0/91 | 0/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Problem Solving Therapy + Behavioral Treatment of Insomnia (N=91) | Enhanced Usual Care (N=90)
Medical or Surgical Hospitalization (Surgical and medical procedures) | 19 (19) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT02145429/Prot_SAP_000.pdf